CLINICAL TRIAL: NCT06323447
Title: Pivotal Study to Validate the Usability, Safety and Diagnostic Performance of a Novel System to Non-Invasively Detect Severe Neutropenia
Brief Title: Pivotal Study to Validate a Novel System to Non-Invasively Detect Severe Neutropenia
Acronym: PC002
Status: Not yet recruiting | Type: Observational
Sponsor: Leuko Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PC002
Record Dates: First submitted 2023-08-21; First posted 2024-03-21 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: PointCheck — Binary classification of severe neutropenia

SUMMARY:
Pivotal study to validate the diagnostic performance of PointCheck, the first non invasive device to preliminary detect neutropenia in cancer patients receiving intermediate/high risk antineoplastic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the purpose and risks of the study and to provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
* Male or Female aged 10 years or above.
* Diagnosed with either Diffuse Large B Cell Lymphoma or Multiple Myeloma.
* Scheduled treatment with any antineoplastic therapy with an associated high/intermediate risk of neutropenia according to NCCN guidelines.
* Able (in the investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Participants with amputations, congenital malformations or any severe abnormalities of the hands as determined by the investigator.
* Participants with a history of vasculitis, Raynaud syndrome, scleroderma, mixed connective tissue disease or any other rheumatologic systemic condition that could produce microcirculatory changes in the nailfold.
* Participants with circulating tumour cells in previous or current lab determinations.
* Participants with any condition producing significant tremor (e.g., essential tremor, Parkinson´s disease, dystonic tremor).
* Unstable participants or participants with hypotension (systolic blood pressure <90 and diastolic blood pressure < 60mmHg).
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrolment.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a multi-site (4 US sites) observational open-label diagnostic study of a non-significant risk medical device, PointCheckTM. Participants (N=210) with specific malignancies who are scheduled to receive antineoplastic therapy will be evaluated during their routine management before the planned cytotoxic drug administration at two-time points (baseline and nadir evaluation). This will be an event-driven study with a total number of 70 positive cases (ANC < 500 cells/mm3) and 140 negative cases (ANC >= 500 cells/mm3) has been considered sufficient to provide accurate estimates of Sensitivity and Specificity. They will have concurrent evaluations with PointCheckTM and a blood differential cell count in addition to the standard clinical visits. A subset (N=45) of patients will be evaluated for between-instrument reproducibility. Finally, a sub-study (N=30) will confirm the usability of PointCheckTM in the home setting.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
PointCheck Accuracy | Two weeks
  The main primary endpoints for this study will be the sensitivity and specificity of PointCheckTM to detect grade IV neutropenia ac cording to the CTCAE V5 definition of severe neutropenia in a standard blood analysis.

SECONDARY OUTCOMES:
PointCheck Precision | Two-weeks
  Repeatability and reproducibility will be assessed using the % positive/negative results of the test's classification compared to the gold standard after multiple measurements in different contexts.
PointCheck Usability | Two-weeks
  Mean System Usability Score
PointCheck Errors | Two-weeks
  Device related errors (number/type)
PointCheck Safety | Two-weeks
  total number (and %) of AEs and SAEs related to the device use.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Castro Gonzalez, PhD, Principal Investigator — Leuko Labs

IPD SHARING:
Plan to Share IPD: Undecided